CLINICAL TRIAL: NCT00546936
Title: Ranibizumab vs PDT for Presumed Ocular Histoplasmosis
Brief Title: Ranibizumab Versus PDT for Presumed Ocular Histoplasmosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Barnes Retina Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Kevin Blinder, MD, Barnes Retina Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF4145s
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2009-04-16 (Estimated); Status verified 2009-04

CONDITIONS: Presumed Ocular Histoplasmosis (POHS)
Keywords: Histoplasmosis
MeSH Terms: conditions — Histoplasmosis | interventions — Ranibizumab; Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ranibizumab intravitreal injection (Experimental): 0.5 mg intravitreal injection of ranibizumab
  Interventions: Drug: ranibizumab
- Photodynamic Therapy (Active Comparator): Photodynamic therapy with Visudyne
  Interventions: Drug: verteporfin

INTERVENTIONS:
Drug: ranibizumab — 0.5mg ranibizumab
  Arms: ranibizumab intravitreal injection
Drug: verteporfin — Photodynamic therapy with verteporfin every 3 months for 1 year
  Other Names: Visudyne
  Arms: Photodynamic Therapy

SUMMARY:
The purpose of this study is to evaluate the change in visual activity of ranibizumab to Photodynamic Therapy (PDT)in patients with choroidal neovascularization (CNV) secondary to presumed ocular histoplasmosis

ELIGIBILITY:
Inclusion Criteria:

* Subfoveal CNV due to presumed ocular histoplasmosis of less than 1 year duration
* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age greater than or equal to 21 years of age
* CNV lesion of than < 5400 microns in diameter
* Best corrected visual acuity of 20/40-20/320
* Birth control therapy for females of child-bearing potential

Exclusion Criteria:

* Subfoveal NCV due tp presumed ocular histoplasmosis for > 1 year
* Pregnancy or lactation premenopausal women not using adequate contraception
* Prior enrollment in the study
* Any other condition that the Investigator believes would pose a significant hazard to the subject
* Participation in another simultaneous medical investigation or trial
* Participation in another trial or previous trial of ranibizumab or Avastin
* Any concurrent ocular condition in the study eye (cataract, diabetic retinopathy)that could require medical or surgical intervention or ifa allowed to progress, could likely contribute to loss of at least 2 Snellen equivalent lines of BCVA over the 12-month study period
* Previous panretinal photocoagulation
* Previous steroids or PDT in 3 months
* Previous participation in any studies of investigational drugs within 30 days preceding Day 0
* Prior participation in a Genentech ranibizumab clinical trial
* Previous treatment with intravitreally (in either eye) or intravenously administered Avastin within 3 months
* Previous use of Macugen in the study eye within 3 months
* Prior submacular surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-10 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Mean change in visual acuity | 6 months, 1 year

SECONDARY OUTCOMES:
To evaluate mean change in vision at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J. Blinder, MD, Principal Investigator — Barnes Retina Institute
Locations (2):
- United States (2):
  - Macula-Retina-Vitreous Service, Midwest Eye Institute, Indianapolis, Indiana
  - Barnes Retina Institute, St Louis, Missouri

REFERENCES:
- [Derived] Ramaiya KJ, Blinder KJ, Ciulla T, Cooper B, Shah GK. Ranibizumab versus photodynamic therapy for presumed ocular histoplasmosis syndrome. Ophthalmic Surg Lasers Imaging Retina. 2013 Jan-Feb;44(1):17-21. doi: 10.3928/23258160-20121221-07. PMID 23410808